CLINICAL TRIAL: NCT00517101
Title: Presence of IBD Specific Antibodies (ASCA, ALCA, ACCA, AMCA) in the Sera of Patients With Spondyloarthropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TAMSC-07-VA-318-CTIL
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: Psoriatic Arthritis; Ankylosing Spondylitis; Undifferentiated Spondyloarthropathy
Keywords: spondyloarthropathy; inflammatory bowel disease; antibodies
MeSH Terms: conditions — Arthritis, Psoriatic; Spondylitis, Ankylosing; Spondylarthropathies; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A relationship between IBD and spondyloarthropathy is well recognized. ASCA ( anti saccharomyces cerevisiae antibodies)are considered to be a serological marker for Crohn's disease and have been studied in patients with spondyloarthropathy with conflicting results. More recently, new serological markers for IBD have been described. These markers are antibodies to certain defined glycans , and their use may permit an improved diagnosis of IBD.

The aim of our study is to investigate wether these new serological markers are present in the sera of patients with spondyloarthropathy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of psoriatic arthritis, ankylosing spondylitis, or undifferentiated spondyloarthropathy

Exclusion Criteria:

* diagnosed inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2007-09

CONTACTS AND LOCATIONS:
Overall Officials: valerie aloush, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center